CLINICAL TRIAL: NCT04646941
Title: Diabetic Complications and Obstructive Sleep Apnea in Type 2 Diabetic Patients: A Longitudinal Study
Brief Title: Diabetic Complications and Obstructive Sleep Apnea
Acronym: DMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-025
Record Dates: First submitted 2020-09-02; First posted 2020-11-30 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Complications and Obstructive Sleep Apnea
Keywords: Type 2 diabetes; diabetic complications; Obstructive Sleep Apnea
MeSH Terms: conditions — Diabetes Complications; Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM with OSA: Type 2 diabetes patients with obstructive sleep apnea
  Interventions: Other: regular treatment
- T2DM without OSA: Type 2 diabetes patients without obstructive sleep apnea
  Interventions: Other: regular treatment

INTERVENTIONS:
Other: regular treatment — The patients with or without OSA received regular hypoglycemic drugs.

SUMMARY:
To follow up the progress of chronic complications in T2DM patients who had undergone anthropometric measurements, laboratory testing and standard overnight polysomnography monitor from 2013 to 2018.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common chronic sleep disorder and a frequent comorbidity in patients with type 2 diabetes. There has been increasing recognition that OSA is highly prevalent in persons with type 2 diabetes. This study is to explore the relationship between OSA and the progress of chronic diabetes-related complications in type 2 diabetes who had undergone anthropometric measurements, laboratory testing and standard overnight polysomnography monitor from 2013 to 2018 in the Department of Endocrinology and Diabetes, The First Affiliated Hospital of Xiamen University, Xiamen, China.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age：18-80

Exclusion Criteria:

* Patients with non type 2 diabetes mellitus
* Preparation for pregnancy
* Lactation patients
* Patients with uncontrolled thyroid disease
* Patients with severe cardiovascular disease
* Patients with severe hepatic and renal insufficiency
* Patients with oral and maxillofacial malformations and upper respiratory tract malformations
* Patients with pulmonary infection or COPD
* Patients who are not willing to accept the questionnaire survey
* Unable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
the progress of diabetic complications | From January 1, 2013 to December 31, 2020
  Diabetic complications include diabetic microvascular complications, atherosclerotic cardiovascular disease(ASCVD), and Diabetic foot disease.
  Diabetic microvascular complications include diabetic nephropathy, diabetic retinopathy and diabetic neuropathy.
  Diabetic macrovascular complications refer to ASCVD, which is defined as coronary heart disease (CHD; acute and silent MI, and unstable angina), ischemic stroke, or peripheral artery disease (PAD).
the new onset and types of tumor in T2DM patients | From January 1, 2013 to December 31, 2020
  the new onset and types of tumor in T2DM patients

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed in this cohort are available from the corresponding author on reasonable request.